CLINICAL TRIAL: NCT01927835
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Homologous and Heterologous Prime-Boost Regimens Comprising DNA-HIV-PT123, NYVAC-HIV-PT1 and NYVAC-HIV-PT4, and AIDSVAX B/E in Healthy, HIV-Uninfected US and South African Adults
Brief Title: Evaluating the Safety and Immune Response to Two HIV Vaccine Regimens in Healthy, HIV-Uninfected Adults in the United States and South Africa
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); IPPOX Foundation (Other); EuroVacc Foundation (Other); Global Solutions for Infectious Diseases (GSID) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 101; 11933 (Registry Identifier: DAIDS-ES ID)
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1A: Treatment (Experimental): Participants will receive the DNA-HIV-PT123 vaccine administered as 1 mL intramuscularly (IM) and placebo (sodium chloride for injection, 0.9%) administered as 1 mL each in the left deltoid at Months 0 and 1. They will then receive the NYVAC-HIV-PT1 vaccine and the NYVAC-HIV-PT4 vaccine; each will be administered as 1 mL IM in the left deltoid and the AIDSVAX B/E vaccine administered as 1 mL IM in the right deltoid at Months 3 and 6.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: NYVAC-HIV-PT1 vaccine; Biological: NYVAC-HIV-PT4 vaccine; Biological: AIDSVAX B/E vaccine; Biological: Placebo for DNA/NYVAC/AIDSVAX
- Group 1B: Treatment (Experimental): Participants will receive the DNA-HIV-PT123 vaccine administered as 1 mL intramuscularly (IM) and placebo (sodium chloride for injection, 0.9%) administered as 1 mL each in the left deltoid at Months 0 and 1. They will then receive the NYVAC-HIV-PT1 vaccine and the NYVAC-HIV-PT4 vaccine; each will be administered as 1 mL IM in the left deltoid and the AIDSVAX B/E vaccine administered as 1 mL IM in the right deltoid at Months 3 and 6.
  Interventions: Biological: DNA-HIV-PT123 vaccine; Biological: NYVAC-HIV-PT1 vaccine; Biological: NYVAC-HIV-PT4 vaccine; Biological: AIDSVAX B/E vaccine; Biological: Placebo for DNA/NYVAC/AIDSVAX
- Group 2A: Treatment (Experimental): Participants will receive the NYVAC-HIV-PT1 vaccine and the NYVAC-HIV-PT4 vaccine, each administered as 1 mL IM in the left deltoid at Months 0 and 1. They will then receive the NYVAC-HIV-PT1 vaccine and the NYVAC-HIV-PT4 vaccine; each will be administered as 1 mL IM in the left deltoid, and the AIDSVAX B/E vaccine administered as 1 mL IM in the right deltoid at Months 3 and 6.
  Interventions: Biological: NYVAC-HIV-PT1 vaccine; Biological: NYVAC-HIV-PT4 vaccine; Biological: AIDSVAX B/E vaccine
- Group 2B: Treatment (Experimental): Participants will receive the NYVAC-HIV-PT1 vaccine and the NYVAC-HIV-PT4 vaccine, each administered as 1 mL IM in the left deltoid at Months 0 and 1. They will then receive the NYVAC-HIV-PT1 vaccine and the NYVAC-HIV-PT4 vaccine; each will be administered as 1 mL IM in the left deltoid, and the AIDSVAX B/E vaccine administered as 1 mL IM in the right deltoid at Months 3 and 6.
  Interventions: Biological: NYVAC-HIV-PT1 vaccine; Biological: NYVAC-HIV-PT4 vaccine; Biological: AIDSVAX B/E vaccine
- Group 3A: Placebo (Placebo Comparator): Participants will receive two injections of placebo (sodium chloride for injection, 0.9%) each administered as 1 mL IM in the left deltoid at Months 0 and 1. They will then receive two injections of placebo (sodium chloride for injection, 0.9%) each administered as 1 mL IM in the left deltoid, and 1 injection of placebo (sodium chloride for injection, 0.9%) administered as 1 mL IM in the right deltoid at Months 3 and 6.
  Interventions: Biological: Placebo for DNA/NYVAC/AIDSVAX
- Group 3B: Placebo (Placebo Comparator): Participants will receive two injections of placebo (sodium chloride for injection, 0.9%) each administered as 1 mL IM in the left deltoid at Months 0 and 1. They will then receive two injections of placebo (sodium chloride for injection, 0.9%) each administered as 1 mL IM in the left deltoid, and 1 injection of placebo (sodium chloride for injection, 0.9%) administered as 1 mL IM in the right deltoid at Months 3 and 6.
  Interventions: Biological: Placebo for DNA/NYVAC/AIDSVAX

INTERVENTIONS:
Biological: DNA-HIV-PT123 vaccine — 4 mg of DNA encoding clade C ZM96 Gag and gp140, CN54 Pol-Nef, administered IM
  Arms: Group 1A: Treatment; Group 1B: Treatment
Biological: NYVAC-HIV-PT1 vaccine — ≥ 5x10^6 PFU/ml encoding clade C ZM96 gp140 for a planned maximum dose of 1.2x10^8 PFU/ml; administered IM
  Arms: Group 1A: Treatment; Group 1B: Treatment; Group 2A: Treatment; Group 2B: Treatment
Biological: NYVAC-HIV-PT4 vaccine — ≥ 5x10^6 PFU encoding ZM96 Gag and CN54 Pol-Nef, administered IM for a planned maximum dose of 1.1x10^7 PFU/ml; administered IM
  Arms: Group 1A: Treatment; Group 1B: Treatment; Group 2A: Treatment; Group 2B: Treatment
Biological: AIDSVAX B/E vaccine — 300 mcg of subtype B (MN) HIV gp120 glycoprotein and 300 mcg of subtype E (A244) HIV gp120 glycoprotein absorbed onto 600 mcg of aluminum hydroxide gel adjuvant, administered IM
  Arms: Group 1A: Treatment; Group 1B: Treatment; Group 2A: Treatment; Group 2B: Treatment
Biological: Placebo for DNA/NYVAC/AIDSVAX — Sodium Chloride for injection, 0.9%; administered IM
  Arms: Group 1A: Treatment; Group 1B: Treatment; Group 3A: Placebo; Group 3B: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to two different HIV vaccine regimens in healthy, HIV-uninfected people in the United States and South Africa.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immune response to two different vaccine schedules of a prime with either DNA HIV vaccine (DNA-HIV-PT123), or NYVAC HIV vaccine (NYVAC-HIV-PT1 and NYVAC-HIV-PT4) followed by a boost combination of NYVAC HIV vaccine (PT1 & PT4) and AIDSVAX B/E. Study researchers will also evaluate whether body mass index (BMI) and/or sex impact the immunogenicity of the vaccine regimens in participants from South Africa, and look at regional differences in immunologic responses between United States and South African participants.

The study will enroll 264 healthy, HIV-uninfected people, ages 18-50, in the United States and South Africa.

Participants will be randomly assigned to one of three groups and receive either one of the vaccine regimens or placebo. Participants will receive injections according to their assigned group schedule at study entry (Month 0) and Months 1, 3, and 6.

Participants will remain in the clinic for 30 minutes after receiving the vaccines for observation and monitoring. For 7 days after receiving the vaccines, participants will record their symptoms and report them to study researchers.

Study visits will occur at study entry, and Months 1, 1.5, 3, 3.5, 6, 6.5, 9, and 12. All study visits will include a physical examination, HIV risk reduction counseling, and interviews and/or questionnaires. Select study visits will include urine collection, an electrocardiogram (ECG), blood collection, a pregnancy test for female participants, and HIV testing. At some visits, some participants may also provide samples of cervical fluid, rectal fluid, and/or semen. Study researchers will contact participants by telephone or e-mail once a year for 3 years following the first vaccination for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent before the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by the clinic staff as being at "low risk" for HIV infection
* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female and greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3
* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal (IULN); creatinine less than or equal to 1.1 times the IULN
* Cardiac Troponin T or I (cTnT or cTnI) does not exceed the IULN
* Negative HIV-1 and -2 blood test: U.S. participants must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA). Non-U.S. sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine:

  1. Negative urine glucose, and
  2. Negative or trace urine protein, and
  3. Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Reproductive status: a participant who was born female must agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, or known hyperlipidemia
* Intent to participate in another study of an investigational research agent during the planned duration of this study
* Pregnant or breastfeeding
* HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the HVTN 101 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA or (South Africa) Medicines Control Council (MCC). For participants who have received control/placebo in an experimental vaccine trial, the HVTN 101 PSRT will determine eligibility on a case-by-case basis. For participants who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 101 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease (Not excluded: mild, well-controlled psoriasis)
* Immunodeficiency
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are people with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  1. If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. More information on this criterion can be found in the protocol.
  2. If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, or clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
* Electrocardiogram (ECG) with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, as determined by the contract ECG lab, cardiologist, or study clinician. More information on this criterion can be found in the protocol.
* Participants who have 2 or more of the following cardiac risk factors: (1) participant report of history of elevated blood cholesterol defined as fasting low-density lipoprotein (LDL) greater than 160 mg/dL; (2) first degree relative (e.g., mother, father, brother, or sister) who had coronary artery disease before the age of 50 years); (3) current smoker; or (4) BMI greater than or equal to 35
* Allergy to eggs or egg products
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of severe local and systemic reactogenicity signs and symptoms | Measured within the initial 7-day period following each vaccination visit and followed until resolution
  Including pain, tenderness, maximum severity of pain and/or tenderness, erythema, induration, fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and maximum severity of systemic symptoms
Frequency of adverse events (AEs) | Measured through participants' last study visit at Month 12
  Including by treatment arm, by body system, Medical Dictionary for Regulatory Activities (MedDRA) preferred term, severity, and assessed relationship to study products
Reports of serious adverse events (SAEs) throughout the active surveillance period | Measured through the end of participants' 3-year follow-up period
Measurements of laboratory measures of safety | Measured through participants' last study visit at Month 12
  Including boxplots of white blood cells (WBC), neutrophils, lymphocytes, hemoglobin, platelets, alanine aminotransferase (ALT), and creatinine at baseline and following vaccinations, by treatment arm
Magnitude and breadth of HIV-specific binding antibody responses as assessed by multiplex assay | Measured 2 weeks after the second NYVAC+AIDSVAX B/E boost or final placebo injection
HIV-specific CD4+ and CD8+ T-cell response rates | Measured 2 weeks after the second NYVAC+AIDSVAX B/E boost or final placebo injection
Magnitude of HIV-specific CD4+ and CD8+ T-cell responses | Measured 2 weeks after the second NYVAC+AIDSVAX B/E boost or final placebo injection
Humoral and cellular vaccine responses for each vaccine regimen in South African men with low BMI and with high BMI | Measured through participants' last study visit at Month 12
Humoral and cellular vaccine responses for each vaccine regimen in South African women with low BMI and with high BMI | Measured through participants' last study visit at Month 12
Humoral and cellular responses to DNA prime followed by NYVAC+AIDSVAX B/E in U.S. adults compared to South African adults | Measured through participants' last study visit at Month 12
Humoral and cellular responses to NYVAC prime followed by NYVAC+AIDSVAX B/E boost in U.S. adults compared to South African adults | Measured through participants' last study visit at Month 12

SECONDARY OUTCOMES:
Magnitude and breadth of HIV-specific binding antibody responses as assessed by multiplex assay | Measured 2 weeks after the second NYVAC+AIDSVAX B/E boost or final placebo injection
HIV-specific CD4+ and CD8+ T-cell response rates | Measured 2 weeks after the second NYVAC+AIDSVAX B/E boost or final placebo injection
Magnitude of HIV-specific CD4+ and CD8+ T-cell responses | Measured 2 weeks after the second NYVAC+AIDSVAX B/E boost or final placebo injection
Humoral and cellular vaccine responses to DNA prime with NYVAC+AIDSVAX B/E boosts and NYVAC prime with NYVAC+AIDSVAX B/E boosts regimens in South African women compared to South African men | Measured through participants' last study visit at Month 12
Humoral and cellular responses to DNA prime with NYVAC+AIDSVAX B/E boosts and NYVAC prime with NYVAC+AIDSVAX B/E boosts regimens in South African women | Measured through participants' last study visit at Month 12
Humoral and cellular responses to DNA prime with NYVAC+AIDSVAX B/E boosts and NYVAC prime with NYVAC+AIDSVAX B/E boosts in South African men | Measured through participants' last study visit at Month 12
Humoral and cellular vaccine responses to DNA prime with NYVAC+AIDSVAX B/E boosts and NYVAC prime with NYVAC+AIDSVAX B/E boosts regimens in South African adults with low and with high BMI | Measured through participants' last study visit at Month 12
Humoral and cellular responses to DNA prime with NYVAC+AIDSVAX B/E boosts and NYVAC prime with NYVAC+AIDSVAX B/E boosts in high BMI South African adults | Measured through participants' last study visit at Month 12
Humoral and cellular responses to DNA prime with NYVAC+AIDSVAX B/E boosts and NYVAC prime with NYVAC+AIDSVAX B/E boosts regimens in low BMI South African adults | Measured through participants' last study visit at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Sobieszczyk, Study Chair — Columbia University